CLINICAL TRIAL: NCT03929809
Title: Iowa Cochlear Implant Clinical Research Center Study of SSD Using Med-El Cochlear Implants
Status: Completed | Type: Observational
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Camille Dunn, Assistant Research Professor, University of Iowa
Other Study IDs: 201901735
Record Dates: First submitted 2019-04-22; First posted 2019-04-29 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2020-09

CONDITIONS: Hearing Loss, Unilateral; Hearing Loss, Profound
MeSH Terms: conditions — Hearing Loss, Unilateral; Hearing Loss | interventions — Cochlear Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Adult Single-sided deafness: Adult subjects with unilateral single-sided deafness at least 6 months (to ensure stability of hearing loss), but no greater than 10 years will be implanted with a MED-EL Synchrony Cochlear Implant.
  Interventions: Device: Cochlear Implant

INTERVENTIONS:
Device: Cochlear Implant — adults with unilateral hearing loss who wish to regain bilateral hearing will be implanted with a cochlear implant on their deafened ear.
  Other Names: MED-EL Synchrony

SUMMARY:
The purpose of this study is to understand the speech perception in noise and in quiet and localization benefits in a laboratory setting in listeners that receive a cochlear implant in an ear with severe to profound hearing loss and have normal, or near-normal hearing in the opposite ear. We will also evaluate the functional benefit of restoring hearing to the impaired ear via questionnaires that subjects will be answering while listening in their natural environment.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be adults who utilize English as their primary language.
2. Unilateral severe to profound sensorineural hearing loss for a duration of at least 6 months (to ensure stability of hearing loss), but no greater than 10 years.
3. Contralateral ear with normal, or near-normal, hearing.
4. Poorer ear (ear to be implanted): severe to profound sensorineural hearing loss, defined as pure-tone thresholds 70 dB HL or greater for the frequencies 500, 1000, 2000, 3000, and 4000 Hz with monosyllabic word understanding, as measured using the CNC Word Test at 60 dBA under earphones, less than or equal to 20%
5. Better ear (contralateral ear): normal or near-normal hearing defined as pure-tone thresholds no poorer than 30 dB HL at 250, 500, 1000, 2000, and 3000 Hz and no poorer than 40 dB HL at 4000 Hz with monosyllabic word understanding, as measured using the CNC Word Test at 60 dBA under earphones, of greater than or equal to 85%.
6. Willingness to comply with all study requirements.
7. Patent cochlea and normal cochlear anatomy.

Exclusion Criteria:

1. Medical or psychological conditions that contraindicate undergoing surgery.
2. Ossification or any other cochlear anomaly that might prevent complete insertion of the electrode array.
3. Unrealistic expectations on the part of the candidate and/or candidate's family, regarding the possible benefits, risks, and limitations that are inherent to the surgical procedure(s) and prosthetic devices.
4. Unwillingness or inability of the candidate to comply with all investigational requirements.
5. Active middle ear infection.
6. Tinnitus primary motivation for implantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be adults 18 years of age or older who utilize English as their primary language. These adults will have unilateral severe to profound sensorineural hearing loss in one ear for a duration of at least 6 months (to ensure stability of hearing loss), but no greater than 10 years. The contralateral ear will present with with normal, or near-normal, hearing.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2021-08-18 (Actual)

PRIMARY OUTCOMES:
Change in AzBio Sentences in Noise | Pre-operative baseline, 3, 6, 12 months post-activation
  The percent correct of words from a list of 20 Target AzBio sentences will be played from 0° azimuth. A list of AzBio sentences will be played in multitalker babble which will be presented in three different conditions: 0° azimuth, S0N90, or S0N270°.
Change in Localization | Pre-operative baseline, 3, 6, 12 months post-activation
  Testing with 16 sounds played randomly from 1 of 8 loudspeakers in a 108 degree arc will be completed with non-implanted ear alone and everyday listening condition at 60 dBA. Subjects will be asked to identify which loudspeaker presented the sound. The RMS error in degrees will be calculated. A lower number indicates better localization ability.

CONTACTS AND LOCATIONS:
Overall Officials: Camille Dunn, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No